CLINICAL TRIAL: NCT02154061
Title: Systems Biology of Inactivated Influenza Vaccine (IIV) in Healthy Adults With or Without Use of Broad Spectrum Antibiotics
Brief Title: Systems Biology of Flu Vaccine in Healthy Adults With and Without the Use of Antibiotics
Acronym: VAX-002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nadine Rouphael, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00074239
Record Dates: First submitted 2014-05-29; First posted 2014-06-03 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Influenza
Keywords: Flu Vaccine, Intestinal Microbiome, Antibiotics
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Metronidazole; Neomycin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IIV Flu Vaccine with Antibiotics (Experimental): This arm will receive antibiotics prior and after IIV administration.
  Interventions: Drug: IIV Flu Vaccine; Drug: Metronidazole; Drug: Neomycin; Drug: Vancomycin
- IIV Flu Vaccine (Active Comparator): This arm will not take antibiotics in conjunction with IIV.
  Interventions: Drug: IIV Flu Vaccine

INTERVENTIONS:
Drug: IIV Flu Vaccine — This is an FDA approved and tested Inactivated Flu Vaccine.
  Other Names: Fluzone
Drug: Metronidazole — This is a standard antibiotic
  Other Names: Flagyl
  Arms: IIV Flu Vaccine with Antibiotics
Drug: Neomycin — This is a standard antibiotic.
  Arms: IIV Flu Vaccine with Antibiotics
Drug: Vancomycin — This is a standard antibiotic.
  Other Names: Vancocin
  Arms: IIV Flu Vaccine with Antibiotics

SUMMARY:
The purpose of the study is to better understand how the use of antibiotics changes micro-organisms in the intestines. The change to micro-organisms in the intestines may change the body's vaccine immune response and alter the effectiveness of the IIV (seasonal flu) vaccine.

In particular, the investigators will be looking at certain markers in blood after vaccination with IIV (seasonal flu vaccine) with or without the use of antibiotics before vaccination.

There will be two randomized groups. Group A will start taking antibiotic by mouth 3 days prior to vaccination and continue taking antibiotics the day of vaccination and one day after vaccination for a total of 5 days. Group B will only receive the IIV (seasonal flu vaccine) and will not take any antibiotics.

The investigators hope to enroll 50 subjects at Emory.

DETAILED DESCRIPTION:
We will study using a system biology approach the immune responses to IIV alone vs. IIV with antibiotic administration

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals aged 18-40 years.
2. Able to understand and give informed consent.
3. Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for ≥1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods for 30 days before and 30 days after TIV vaccination

Exclusion Criteria:

* You received blood product within 3 months of enrolling in the study or a live attenuated vaccine within 4 weeks or inactivated vaccines within 2 weeks.
* You received the 2014-2015 flu vaccine or had a confirmed case of influenza during 2014-2015.
* You received any antibiotics 6 months prior to enrolling in the study or expect to take antibiotics one month after vaccination.
* You received probiotics or prebiotics 3 months prior before enrolling in the study or expect to take one month after vaccination.
* You received proton pump inhibitors, H2 blocker receptors, or antacids 3 months regularly before enrolling in the study or one month after
* You had an allergic response or sensitivity to past vaccinations.
* You have health conditions that weaken your body's ability to fight infections or you are taking drugs like steroids that weaken your body's ability to fight infections.(Some nasal and topical steroids are allowed.).
* You have a chronic medical problem including (but not limited to) insulin dependent diabetes, severe heart disease including arrhythmias, severe lung disease, auto immune diseases and or grade 4 uncontrolled hypertension.
* Chronic neurological conditions such as seizure disorder, Parkinson disease, myasthenia gravis, neuropathy, or histories of encephalopathy, meningitis or ototoxicity.
* Any history of gastrointestinal disease, kidney or liver diseases.
* Alcohol or drug abuse or psychiatric conditions that in the opinion of the investigator would compromise your participation in this trial.
* Pregnant or are breast feeding.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-04; Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- Emory Vaccine Center, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Wimmers F, Donato M, Kuo A, Ashuach T, Gupta S, Li C, Dvorak M, Foecke MH, Chang SE, Hagan T, De Jong SE, Maecker HT, van der Most R, Cheung P, Cortese M, Bosinger SE, Davis M, Rouphael N, Subramaniam S, Yosef N, Utz PJ, Khatri P, Pulendran B. The single-cell epigenomic and transcriptional landscape of immunity to influenza vaccination. Cell. 2021 Jul 22;184(15):3915-3935.e21. doi: 10.1016/j.cell.2021.05.039. Epub 2021 Jun 25. PMID 34174187

RESULTS

PARTICIPANT FLOW:
Groups:
- IIV Flu Vaccine With Antibiotics: This arm will receive antibiotics prior and after IIV administration.
  Arm 1 and Arm 2: Inactivated Flu Vaccine: This is an FDA approved and tested Flu Vaccine.
  Metronidazole: This is a standard antibiotic
  Neomycin: This is a standard antibiotic.
  Vancomycin: This is a standard antibiotic.
- IIV Flu Vaccine: This arm will not take antibiotics in conjunction with IIV.
  Arm 1 and Arm 2: Inactivated Flu Vaccine: This is an FDA approved and tested Flu Vaccine.
Period: Overall Study
Arm/Group | IIV Flu Vaccine With Antibiotics | IIV Flu Vaccine
Started | 16 | 17
Completed | 14 | 17
Not Completed | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — enrolled but not vaccinated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IIV Flu Vaccine With Antibiotics | IIV Flu Vaccine | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 9 | 8 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 8 | 8 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Four Fold Rise in HAI Titers or HAI 1:40 and Above in Each Group at D30
Description: Number of participants with four fold rise in HAI titers or HAI 1:40 and above in each group at D30 will be recorded based on immunologic testing of blood samples
Time Frame: At day 30
Population: The Overall Number of Participants analyzed for "IIV Flu Vaccine with Antibiotics" is 15, as one participant received antibiotics and did not receive vaccine. The study personnel were unable to draw blood on her at the vaccination day- therefore she was part of the safety population and not the immunogenicity population.
Measure: Count of Participants; unit: Participants
Arm/Group | IIV Flu Vaccine With Antibiotics | IIV Flu Vaccine
Number analyzed (Participants) | 15 | 17
Participants | 15 | 17

ADVERSE EVENTS:
Time Frame: 365 days
Arm/Group | IIV Flu Vaccine With Antibiotics | IIV Flu Vaccine
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 6/16 | 3/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IIV Flu Vaccine With Antibiotics (N=16) | IIV Flu Vaccine (N=17)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (General disorders) | 3 (3) | 0 (0)
anemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
anal itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT02154061/Prot_SAP_000.pdf